CLINICAL TRIAL: NCT06911502
Title: A Phase 3, Multicenter, Randomized, Open Label Study to Compare the Efficacy and Safety of Golcadomide in Combination With Rituximab (Golca + R) Vs Investigator's Choice in Participants With Relapsed/Refractory Follicular Lymphoma Who Have Received at Least 1 Prior Line of Systemic Therapy
Brief Title: A Study to Compare the Efficacy and Safety of Golcadomide in Combination With Rituximab (Golca + R) vs Investigator's Choice in Participants With Relapsed/Refractory Follicular Lymphoma Who Have Received at Least 1 Prior Line of Systemic Therapy (GOLSEEK-4)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA073-1003; 2024-519152-82 (Other: EU CTR); U1111-1314-3909 (Other: WHO)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; Second Line Follicular Lymphoma; Third Line Follicular Lymphoma; Relapsed/refractory follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Lenalidomide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Golcadomide + Rituximab (Experimental)
  Interventions: Drug: Golcadomide; Drug: Rituximab
- Rituximab + Lenalidomide/Chemotherapy (Active Comparator): Rituximab + Lenalidomide or R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone/prednisolone) or Rituximab + Bendamustine
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prednisolone; Drug: Bendamustine

INTERVENTIONS:
Drug: Golcadomide — Specified dose on specified days
  Other Names: CC-99282; BMS-986369
  Arms: Golcadomide + Rituximab
Drug: Rituximab — Specified dose on specified days
Drug: Lenalidomide — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy
Drug: Cyclophosphamide — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy
Drug: Doxorubicin — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy
Drug: Vincristine — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy
Drug: Prednisone/Prednisolone — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy
Drug: Bendamustine — Specified dose on specified days
  Arms: Rituximab + Lenalidomide/Chemotherapy

SUMMARY:
The study is designed as a multicenter, randomized, open label Phase 3 study to compare the efficacy and safety of golcadomide in combination with rituximab vs investigator's choice in participants with relapsed/refractory follicular lymphoma who have received at least one line of prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed FL (Grade 1, 2, 3a or classic FL) as assessed by local pathology. Adequate fresh tumor biopsy tissue or archived tumor biopsy from the latest relapse if available with corresponding pathology report for retrospective central pathology confirmation of relapse, is required. Evaluation from fine needle aspirate is not permitted.
* Relapsed or refractory disease:

  1. Relapsed FL is defined as relapse after an initial response of CR or PR to the most recent prior therapy.
  2. Refractory FL is defined as best response of SD or PD or a response that lasted less than 6 months to the most recent prior therapy.
* Eastern Cooperative Oncology Group (ECOG) 0-2 (ECOG 3 authorized if it is due to lymphoma and not comorbidities).
* Participant must have positron emission tomography (PET)-positive disease with at least one PET-positive lesion and measurable disease on cross section imaging by CT, as defined by Lugano classification.
* Participants with an indication for anti-lymphoma treatment as per investigator assessment based on modified Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria.
* Participant has received at least 1 or more prior lines of systemic therapy with one line consisting of a combination including an anti-CD20 monoclonal antibody (eg, rituximab, obinutuzumab) and an alkylating agent (eg, cyclophosphamide, bendamustine). Prior treatment with radiation therapy does not count as a line of therapy for eligibility.
* Lab parameters:

  1. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 (1.0 x 109 /L),
  2. PLT count ≥ 75,000 cells/mm3 (75 x 109 /L)
  3. Hb ≥ 7.5 g/dL
* estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73m².
* Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤ 2.5 x upper limit of normal (ULN). In case of documented liver involvement by lymphoma, ALT/SGPT and AST/SGOT must be ≤ 5.0× ULN.
* Serum total bilirubin ≤ 1.5 × ULN (corresponding to mild dysfunction as per National Cancer Institute Organ Dysfunction Working Group [NCI ODWG] criteria). In case of documented liver involvement by lymphoma, serum total bilirubin must be ≤ 3.0 × ULN (corresponding to moderate dysfunction as per NCI ODWG criteria). For cases of Gilberts syndrome, serum total bilirubin≤ 5.0 × ULN
* Adequate cardiac function for participants receiving anthracycline-based chemotherapy, defined as left ventricular ejection fraction (LVEF) ≥ 45% as assessed by echocardiogram (ECHO) as standard of care or multi-gated acquisition scan (MUGA)

Exclusion Criteria:

* Evidence or history of composite Diffuse large B-cell lymphoma (DLBCL) and FL or of transformed Non-Hodgkin Lymphoma (NHL) or any other indolent lymphoma.
* Follicular large cell as per 5th World Health Organization (WHO) sub-classification (grade 3b FL per WHO 4th classification) or duodenal-type FL.
* Participant has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from compliantly participating in the study based on Investigator's judgment.
* Participant has any condition that confounds the ability to interpret data from the study based on Investigator's or Sponsor's judgment.
* Presence or history of central nervous system (CNS) involvement by lymphoma.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Deep venous thrombosis/Pulmonary embolism within 1 month prior to enrollment.
* Participants with a history of progressive multifocal leukoencephalopathy.
* Participant has any other subtype of lymphoma.
* Participant has persistent diarrhea or malabsorption ≥ Grade 2 (NCI CTCAE v5.0), despite medical management.
* History of another primary malignancy that has not been in remission for ≥ 3 years except for non-invasive malignancies.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-04-24 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by Independent Review Adjudication committee (IRAC) | Up to approximately 32 Months

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by IRAC | Up to approximately 32 Months
Overall survival (OS) | Up to approximately 83 Months
PFS as assessed by investigator | Up to approximately 32 Months
ORR as assessed by investigator | Up to approximately 32 Months
Number of participants who achieve complete metabolic response (CMR) | Up to approximately 32 Months
Duration of Response (DoR) | Up to approximately 32 Months
Event free survival (EFS) | Up to approximately 32 Months
Time to next anti-lymphoma treatment (TTNT) | Up to approximately 32 Months
PFS on next anti-lymphoma treatment (PFS2) | Up to approximately 32 Months
Time from randomization to meaningful improvement in primary domains of interest in the European Organization for Research and Treatment of Cancer - Quality of Life C30 (EORTC QLQ-C30) Questionnaire | Up to approximately 32 Months
Time from randomization to meaningful improvement in primary domains of interest in the European Organization for Research and Treatment of Cancer - Non- Hodgkin Lymphoma- Low Grade- 20 items (EORTC QLQNHL- LG20) Questionnaire | Up to approximately 32 Months
Minimal residual disease (MRD) negativity | Up to approximately 32 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (160):
- United States (31):
  - Local Institution - 0225, Birmingham, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Local Institution - 0215, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Local Institution - 0008, Jacksonville, Florida
  - Local Institution - 0214, Tampa, Florida
  - Local Institution - 0217, Tampa, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Local Institution - 0240, Arlington Heights, Illinois
  - Local Institution - 0253, Iowa City, Iowa
  - Local Institution - 0243, Waukee, Iowa
  - Local Institution - 0216, Westwood, Kansas
  - Local Institution - 0218, Lexington, Kentucky
  - Local Institution - 0023, Baltimore, Maryland
  - Greater Baltimore Medical Center, Towson, Maryland
  - Local Institution - 0145, Boston, Massachusetts
  - Local Institution - 0244, Boston, Massachusetts
  - Local Institution - 0247, Boston, Massachusetts
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Local Institution - 0144, Providence, Rhode Island
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Local Institution - 0212, Fort Worth, Texas
  - Local Institution - 0230, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Local Institution - 0238, Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Local Institution - 0143, Vancouver, Washington
- Australia (7):
  - Westmead Hospital, Westmead, New South Wales
  - Local Institution - 0132, Adelaide, South Australia
  - Local Institution - 0131, Hobart, Tasmania
  - Local Institution - 0128, Heidelberg, Victoria
  - Cabrini Hospital - Malvern, Malvern, Victoria
  - Local Institution - 0127, Perth, Western Australia
  - Local Institution - 0224, Perth, Western Australia
- Brazil (7):
  - Local Institution - 0159, Vitória, Espírito Santo
  - Local Institution - 0088, Niterói, Rio de Janeiro
  - Local Institution - 0087, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0079, São Paulo, São Paulo
  - Local Institution - 0089, Rio de Janeiro
  - Local Institution - 0066, São Paulo
  - Local Institution - 0092, São Paulo
- Canada (5):
  - Local Institution - 0200, Victoria, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Local Institution - 0250, Québec, Quebec
  - Local Institution - 0192, Sherbrooke, Quebec
  - Local Institution - 0226, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0154, Santiago, Santiago Metropolitan
  - Local Institution - 0155, Santiago, Santiago Metropolitan
  - Local Institution - 0153, Santiago, Santiago Metropolitan
- China (23):
  - Local Institution - 0246, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Local Institution - 0172, Fuzhou Fujian, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Local Institution - 0241, Harbin, Heilongjiang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Local Institution - 0175, Changsha, Hunan
  - Inner Mongolia Cancer Hospital, Hohhot, Inner Mongolia
  - Local Institution - 0233, Suzhou, Jiangsu
  - Local Institution - 0178, Nanchang, Jiangxi
  - Local Institution - 0239, Changchun, Jilin
  - Local Institution - 0177, Changchun, Jilin
  - Local Institution - 0179, Shenyang, Liaoning
  - Local Institution - 0242, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Local Institution - 0181, Shanghai, Shanghai Municipality
  - Local Institution - 0249, Shanghai, Shanghai Municipality
  - Local Institution - 0234, Sichuan, Sichuan
  - Local Institution - 0182, Tianjin, Tianjin Municipality
  - Tianjin People' s Hospital, Tianjin, Tianjin Municipality
  - Local Institution - 0248, Kunming, Yunnan
  - Local Institution - 0184, Hangzhou, Zhejiang
  - Local Institution - 0174, Zhengzhou
- Finland (3):
  - Local Institution - 0151, Oulu, North Ostrobothnia
  - Local Institution - 0152, Turku, Southwest Finland
  - Local Institution - 0150, Helsinki
- France (8):
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Local Institution - 0044, Saint-Cloud, Hauts-de-Seine
  - Chu Saint Eloi, Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Loire-Atlantique
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Local Institution - 0042, Pierre-Bénite, Rhône
  - Local Institution - 0191, Paris
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse
- Germany (14):
  - Local Institution - 0163, Ulm, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Local Institution - 0220, Göttingen, Lower Saxony
  - GEFOS Gesellschaft f. onkologische Studien, Dortmund, North Rhine-Westphalia
  - Local Institution - 0193, Düsseldorf, North Rhine-Westphalia
  - Local Institution - 0231, Münster, North Rhine-Westphalia
  - Local Institution - 0232, Münster, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes, Homburg, Saarland
  - HELIOS Klinikum Erfurt, Erfurt, Thuringia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Klinikum Chemnitz Ggmbh, Chemnitz
  - Gemeinschaftspraxis Hämatologie - Onkologie Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Local Institution - 0162, München
  - Local Institution - 0221, Würzburg
- Greece (6):
  - Local Institution - 0111, Alexandroupoli, Anatolikí Makedonía Kai Thráki
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - General Hospital of Athens "Laiko", Αthens, Attikí
  - Local Institution - 0110, Thessaloniki, Thessaloníki
  - Local Institution - 0197, Thessaloniki, Thessaloníki
  - Local Institution - 0108, Ioannina, Ípeiros
- India (5):
  - Local Institution - 0139, Bengaluru, Karnataka
  - Local Institution - 0141, Mumbai, Maharashtra
  - Local Institution - 0142, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0140, Hyderabad, Telangana
  - Local Institution - 0138, Hyderabad, Telangana
- Italy (7):
  - Local Institution - 0104, Bologna, Emilia-Romagna
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Local Institution - 0102, Alessandria
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Local Institution - 0157, Torino
- Japan (10):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Aiiku Hospital, Sapporo, Hokkaido
  - Japanease Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashiku, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
- Netherlands (3):
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
  - Local Institution - 0046, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (5):
  - AIDPORT Sp. z o.o., Skórzewo, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Local Institution - 0190, Gdynia, Pomeranian Voivodeship
  - Local Institution - 0189, Lodz, Łódź Voivodeship
- Saudi Arabia (3):
  - Local Institution - 0099, Dammam, Eastern Province
  - Local Institution - 0054, Riyadh
  - Local Institution - 0052, Riyadh
- South Korea (4):
  - Local Institution - 0059, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0060, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0061, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0058, Seoul
- Spain (6):
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona [Barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Infanta Leonor, Madrid, Madrid, Comunidad de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Virgen Nieves, Granada
  - Local Institution - 0123, Madrid
- Turkey (Türkiye) (4):
  - Local Institution - 0195, Istanbul- Fatih, Istanbul
  - Local Institution - 0194, Ankara
  - Local Institution - 0196, Antalya
  - Local Institution - 0223, Mersin
- United Arab Emirates (2):
  - Local Institution - 0251, Abu Dhabi, Abu Dhabi Emirate
  - Local Institution - 0252, Abu Dhabi, Abu Dhabi Emirate
- United Kingdom (4):
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Cringleford, England
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Local Institution - 0213, London, London, City of
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06911502.html